CLINICAL TRIAL: NCT06151405
Title: Individualized Nutrition to Help Asthmatics Improve Lung Function and Energetics (INHALE)
Brief Title: Nutrition for Asthmatics
Acronym: INHALE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jacob T. Mey, PhD RD, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBRC 2022-001 B; 1K01HL169491-01 (NIH)
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Asthma
Keywords: ketone; diet; metabolism
MeSH Terms: conditions — Asthma; Ketosis | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not be made aware of the diet allocation. However, due inherent differences in macronutrient content of the diets, participants may perceive differences in the quantity of various food groups or in the taste, texture or smell of foods present in the diet. To address this, diets will be designed to minimize noticeable differences for the participant. The investigator and outcomes assessor will remain fully masked to diet provision.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary Guidelines for Americans (Experimental): 7 days of a diet consistent with the Dietary Guidelines for Americans (DGA).
  Interventions: Other: DGA Diet
- Medium Chain Triglyceride Supplemented DGA (Experimental): 7 days of a diet consistent with the Dietary Guidelines for Americans supplemented with medium chain triglycerides (MCT).
  Interventions: Other: MCT Diet
- Ketogenic Diet (Experimental): 7 days of a ketogenic diet (KETO).
  Interventions: Other: KETO Diet

INTERVENTIONS:
Other: DGA Diet — A fully provisioned isocaloric, isonitrogenous study diet following the Dietary Guidelines for Americans (DGA)
  Including:
  * A variety of vegetables and fruits
  * Grains, at least half of which are whole grains
  * Fat-free or low-fat dairy
  * A variety of protein foods, including seafood, lean meats and poultry, eggs, legumes, nuts, and seeds
  * This healthy eating pattern also limits saturated fats and trans fats, added sugars, and sodium.
  Arms: Dietary Guidelines for Americans
Other: MCT Diet — A fully provisioned isocaloric, isonitrogenous study diet following the Dietary Guidelines for Americans supplemented with medium chain triglycerides (MCT).
  Arms: Medium Chain Triglyceride Supplemented DGA
Other: KETO Diet — A fully provisioned isocaloric, isonitrogenous ketogenic study diet.
  Arms: Ketogenic Diet

SUMMARY:
Determine to what extent three distinct dietary approaches improve asthma control and lung function.

DETAILED DESCRIPTION:
This is a crossover design pilot trial that will recruit 15 adults with asthma. Participants will undergo screening and a lead-in period before being randomized to a series of three, 7-day diets with a 7+ day washout period between each diet. Asthma control and lung function will be assessed at the completion of each diet.

The goal of this pilot trial is to understand the effect of diet on asthma and conduct an exploratory analysis on factors that may predict the response to diet.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* BMI: 18.5 - 29.99 kg/m2
* asthma diagnosed by medical specialist (confirmed in medical history)
* partly controlled or uncontrolled asthma by Asthma Control Test score ≤22
* owns a device compatible with ZEPHYRx platform
* stable asthma medication use (no change in the past 2 months).

Exclusion Criteria:

* Diabetes or using diabetes medications that may lower blood glucose levels
* point of care fasting blood glucose ≥126 mg/dl or triglycerides ≥400 mg/dl
* current smoking or smoking history of greater than 10 pack-years
* other significant respiratory or cardiac disease or the presence of clinically important comorbidities, e.g., COPD, renal failure, liver disease; uncontrolled hypertension defined as systolic blood pressure ≥160 mm/Hg, or diastolic blood pressure ≥100 mm/Hg
* pregnant or nursing women
* food preferences or allergies inconsistent with study diet capabilities
* noncompliance with lead-in period requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Asthma Control | Baseline
  Asthma Control Questionnaire score (Juniper; 1 week recall period) Score range: 0-6. Minimally important difference = 0.5.
Asthma Control | After 7 days on Diet#1
  Asthma Control Questionnaire score (Juniper; 1 week recall period) Score range: 0-6. Minimally important difference = 0.5.
Asthma Control | After 7 days on Diet#2
  Asthma Control Questionnaire score (Juniper; 1 week recall period) Score range: 0-6. Minimally important difference = 0.5.
Asthma Control | After 7 days on Diet#3
  Asthma Control Questionnaire score (Juniper; 1 week recall period) Score range: 0-6. Minimally important difference = 0.5.
Lung Function | Baseline
  FEV1 (forced expiratory volume in 1 second; % of predicted)
Lung Function | After 7 days on Diet#1
  FEV1 (forced expiratory volume in 1 second; % of predicted)
Lung Function | After 7 days on Diet#2
  FEV1 (forced expiratory volume in 1 second; % of predicted)
Lung Function | After 7 days on Diet#3
  FEV1 (forced expiratory volume in 1 second; % of predicted)

SECONDARY OUTCOMES:
Systemic inflammation | Baseline
  plasma interleukin-6 (IL6)
Systemic inflammation | After 7 days on Diet#1
  plasma interleukin-6 (IL6)
Systemic inflammation | After 7 days on Diet#2
  plasma interleukin-6 (IL6)
Systemic inflammation | After 7 days on Diet#3
  plasma interleukin-6 (IL6)
FENO | Baseline
  FENO (ppm)
FENO | After 7 days on Diet#1
  FENO (ppm)
FENO | After 7 days on Diet#2
  FENO (ppm)
FENO | After 7 days on Diet#3
  FENO (ppm)
FEV1/FVC | Baseline
  FEV1/Forced Vital Capacity (FVC) ratio
FEV1/FVC | After 7 days on Diet#1
  FEV1/Forced Vital Capacity (FVC) ratio
FEV1/FVC | After 7 days on Diet#2
  FEV1/Forced Vital Capacity (FVC) ratio
FEV1/FVC | After 7 days on Diet#3
  FEV1/Forced Vital Capacity (FVC) ratio

OTHER OUTCOMES:
indirect calorimetry | baseline, after 7 days on Diet#1, after 7 days on Diet#2, after 7 days on Diet#3
  nutrient utilization according to respiratory exchange ratio (0.66 - 1.0)
ketosis | baseline, after 7 days on Diet#1, after 7 days on Diet#2, after 7 days on Diet#3
  plasma ß-hydroxybutyrate (mM)
eosinophilic asthma characterization | baseline, after 7 days on Diet#1, after 7 days on Diet#2, after 7 days on Diet#3
  absolute blood eosinophils (count)
immunoglobulin asthma characterization | baseline, after 7 days on Diet#1, after 7 days on Diet#2, after 7 days on Diet#3
  blood immunoglobulin E (IgE)
systemic inflammation | baseline, after 7 days on Diet#1, after 7 days on Diet#2, after 7 days on Diet#3
  blood cytokines (IL17, TNFα, IL1ß)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Mey, PhD, RD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
IPD is stored according to our institutional policy. External investigators may request additional data access, which will be shared according to institutional policy with appropriate data sharing agreements.